CLINICAL TRIAL: NCT05696977
Title: Effect of Obesity on Cyclosporine Blood Trough Level in Nephrotic Syndrome Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107113
Record Dates: First submitted 2022-12-15; First posted 2023-01-25 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Nephrotic Syndrome
Keywords: Cyclosporine; Obese patients; Lipoproteins
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: Open labelled, prospective,non-randomized, two-arms,parallel groups, non-placebo controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obese nephrotic patients with BMI>25 kg/m2 (Active Comparator): Nephrotic obese patients receive Cyclosporine capsule initially according to weight-based dose then modifying the dose according to targeted therapeutic level.
  To determine the best weight can be used to get the targeted therapeutic level. Correlate with the lipid profile, fat percentage and other anthropometric measures.
  Interventions: Drug: Cyclosporine Capsule
- Non obese nephrotic patients with BMI<25 kg/m2 (Other): Nephrotic non-obese patients receive Cyclosporine capsule initially according to weight-based dose then modified dose according to targeted therapeutic level.
  Interventions: Drug: Cyclosporine Capsule

INTERVENTIONS:
Drug: Cyclosporine Capsule — Determination of the most appropriate weight based dose of Cyclosporine to achieve the target therapeutic drug level and response and its relation with fat percentage and lipid profile

SUMMARY:
This study aims to assess the effect of obesity on therapeutic response and safety of cyclosporine trough level in nephrotic syndrome patients and calculating a suitable weight-based dose.

DETAILED DESCRIPTION:
1. Ethical committee approval has been obtained from Ethics committee of Faculty of Medicine, Alexandria University.
2. Agreement from all participants should be taken in this clinical study by assigning an informed consent.
3. Nephrotic diseased patients,will be recruited from Alexandria main university hospital (AMUH).
4. The 74 participants will be non-randomly assigned into 2 groups.
5. The control group is non-obese nephrotic patients with BMI <25 kg/m2 will receive receive Cyclosporine capsule with conventional initial dose 3 mg/kg/day using actual weight.
6. The Case interventional group is Obese nephrotic patients with BMI> 25kg/m2 will receive Cyclosporine capsule with the best weight based dose to achieve the targeted therapeutic trough level and targeted urinary protein/ creatinine ratio.
7. All patients will be subjected to :

   * First visit: Full patient history, anthropometrics (weight, hight, BMI, fat %, water %, muscles% and clinical examination. Calculate the initial cyclosporine dose 3mg/kg/day in 2 divided doses based on actual weight.
   * Second visit after one month: blood sample withdrawal for measuring trough level, lipid profile and thyroid profile, urinary sample to measure uPCR If patients don't reach to targeted therapeutic trough level and targeted urinary protein/ creatinine ratio,re-modifying the dose and repeat the labs after another one month in third visit.
   * Finally find the best weight can be used to achieve the targeted therapeutic trough level and targeted urinary protein/ creatinine ratio, and its relation with fat content and lipid profile
8. The appropriate Statistical tests will be hold according to study design and parameters (parametric and non-parametric) to evaluate the significance of the results.
9. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Obese and overweight Nephrotic syndrome adult patients receiving Cyclosporine for more than one month with prednisolone. (BMI>25 kg/m2)
* Normal or underweight individuals Nephrotic syndrome adult patients receiving Cyclosporine for more than one month with prednisolone. (serving as control group)

Exclusion Criteria:

* Hepatic patients liver cirrhosis (moderate to severe liver impairment)
* Cancer patients,
* Pregnant and lactating female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-04-17 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Cyclosporine level concentration and its correlation to anthropometric measures | 1 month
  Measuring of Cyclosporine level in whole blood after one month of starting the drug
Determine a suitable weight-based dose for obese patients | 1 month
  Modifying the Cyclosporine dose according to measured trough level
Measuring the weight as one of anthropometric measures | Day 1
  Measuring anthropometric measures as; weight in kilograms at base line of starting the Cyclosporine regimen.
Measuring the height as one of anthropometric measures | Day 1
  Measuring anthropometric measures as;height in metres at base line of starting the Cyclosporine regimen.
Measuring the BMI as one of anthropometric measures | Day 1
  Measuring anthropometric measures as; BMI (body mass index) in kilograms/meter^2 at base line of starting the Cyclosporine regimen.
Measuring some of important in-body anthropometric measures | Day 1
  Measuring anthropometric measures as;body fat percentage, body water percentage and muscle percentage content at base line of starting the Cyclosporine regimen.

SECONDARY OUTCOMES:
Assessment of kidney functions | 1 month
  Measuring parameters represent the kidney functions including (serum creatinine in mg/dl.)
Assessment of kidney functions as clearance estimation | 1 month
  Measuring parameters represent the kidney functions including (estimated GFR in mL/min/1.73 m²)
Assessment of kidney functions as urinary protein release | 1 month
  Measuring parameters represent the kidney functions including (Urinary protein-creatinine ratio in gm/gm)
Lipid profile assessment | 1 month
  Measuring lipid profile including (HDL, LDL,VLDL and TG) in mg/dl.
Thyroid function assessment | 1 month
  Measuring Thyroid profile including (TSH, fT3, fT4 ).
Covid-19 vaccine status assessment | Day 1
  Assess if the patient received Covid-19 vaccine, or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No